CLINICAL TRIAL: NCT06889259
Title: Efficacy and Safety of Cognitive Behavioral Therapy, Tones Stimulator in Patients With Subjective Tinnitus: Prospective, Multi-center, Randomized, Single Blind (Subject), Parallel, Superiority, Confirmatory Trial
Brief Title: Efficacy and Safety of CBT on Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023GR0400
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-center, Randomized, single blind (subject), Parallel, Superiority, Confirmatory Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT based digital therapeutics (Active Comparator): CBT using digital therapeutics
  Interventions: Behavioral: CBT based digital therapeutics
- Conventional CBT (Sham Comparator): Conventional CBT
  Interventions: Behavioral: Conventional CBT

INTERVENTIONS:
Behavioral: CBT based digital therapeutics — The mobile-based digital therapeutic intervention integrated video education, thought record sheets, and sound therapy. This comprehensive treatment was administered five times weekly. The program consisted of a total of 30 sessions.
  Arms: CBT based digital therapeutics
Behavioral: Conventional CBT — The cognitive behavioral therapy program for tinnitus, based on a paper manual, was administered five times per week. The treatment regimen consisted of a total of 30 sessions,.
  Arms: Conventional CBT

SUMMARY:
Tinnitus, the perception of sound without external stimuli, affects 14% of the global population, posing a significant public health concern. This predominantly subjective condition often leads to psychological and physical distress, including anxiety, depression, and insomnia. As tinnitus prevalence rises due to aging populations and increased noise exposure, the need for effective treatments grows urgent.

Current approaches include pharmacological interventions, sound therapy, and cognitive behavioral therapy (CBT), with CBT recognized as most effective for addressing psychological distress. However, traditional therapies face accessibility barriers such as frequent in-person sessions and high costs.

Digital therapeutics, particularly mobile applications, offer promising solutions by providing scalable, accessible interventions. These allow patients to engage in therapy conveniently, accessing real-time, personalized content. Despite advancements, research on digital therapeutics combining CBT and sound therapy for tinnitus remains limited.

This study aims to address this gap by evaluating the clinical efficacy of a mobile application delivering personalized CBT and sound stimulation compared to conventional CBT, potentially contributing to more accessible and effective tinnitus treatment options.

DETAILED DESCRIPTION:
Tinnitus, characterized by the perception of sound without external stimuli, affects approximately 14% of the global population, posing a significant public health concern. This predominantly subjective condition often leads to psychological and physical distress, including anxiety, depression, and insomnia. Current approaches to managing tinnitus include pharmacological interventions, sound therapy, and cognitive behavioral therapy (CBT). Among these, CBT is recognized as one of the most effective methods for addressing the psychological distress associated with tinnitus. However, traditional CBT often faces accessibility barriers, such as the need for frequent in-person sessions and high costs. This limits its reach and effectiveness for many patients.Digital therapeutics, particularly mobile applications, offer promising solutions by providing scalable and accessible interventions. These platforms allow patients to engage in therapy conveniently, accessing real-time, personalized content. Despite advancements in digital therapeutics, research on combining CBT and sound therapy for tinnitus remains limited. This gap in research highlights the need for innovative, accessible treatments that can be tailored to individual patient needs.

This study aims to address this gap by evaluating the clinical efficacy of a mobile application that delivers personalized CBT and sound stimulation. The application, designed to provide tailored interventions, will be compared to conventional CBT methods. By leveraging the strengths of both CBT and sound therapy, this study seeks to contribute to the development of more accessible and effective tinnitus treatment options.

The study will employ a prospective, multicenter, randomized, single-blind (participant), parallel-design, superiority, confirmatory trial to assess the efficacy and safety of the mobile application. Participants will be randomly assigned to either the intervention group using the mobile application or the control group receiving conventional CBT educational materials. The primary outcome will be the change in Tinnitus Handicap Inventory (THI) scores from baseline to 6 weeks, with secondary outcomes including changes in THI subscales, Tinnitus Functional Index (TFI), Visual Analog Scale (VAS) for negative emotions and tinnitus discomfort, Beck Depression Inventory (BDI), and Beck Anxiety Inventory (BAI).

The study's design and methodology are crucial for evaluating the effectiveness of the mobile application. By using a randomized controlled trial design, the study ensures that any observed effects can be attributed to the intervention rather than external factors. The use of standardized assessment tools like THI and TFI will provide a comprehensive understanding of the application's impact on tinnitus-related distress.

Furthermore, the study will assess the safety and tolerability of the mobile application, monitoring for any adverse events or side effects. This is essential for ensuring that the treatment is not only effective but also safe for widespread use.

ELIGIBILITY:
Inclusion Criteria:

* Subjective tinnitus more than 3mo
* age over 19
* Pure tone audiometry < 60 decibel
* Tinnitus handicap inventory score > 18

Exclusion Criteria:

* Objective tinnitus
* Otitis, labyrinthitis
* Depression, Anxiety, Insomnia or other psychiatric disorder
* Pregnancy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Tinnitus handicap inventory | Baseline, 4weeks, 5weeks 6weeks
  The Tinnitus Handicap Inventory is a widely used 25-item self-report questionnaire designed to assess the impact of tinnitus on an individual's daily life. It evaluates functional, emotional, and catastrophic effects of tinnitus, with scores ranging from 0 to 100. Higher score means worse outcome。

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Jun Song, Study Director — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT06889259/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT06889259/ICF_001.pdf